CLINICAL TRIAL: NCT03920163
Title: Enhanced Recovery After Trauma Surgery
Acronym: ERATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Dr DEK McPherson, Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERATS
Record Dates: First submitted 2019-04-05; First posted 2019-04-18 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Penetrating Abdominal Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Stable , penetrating trauma patients undergoing laparotomy who receive standard post operative care
  Interventions: Other: Enhanced Recovery Measures
- ERATS (Experimental): Stable penetrating trauma patients undergoing laparotomy who receive enhanced recovery measures post operatively .
  Interventions: Other: Enhanced Recovery Measures

INTERVENTIONS:
Other: Enhanced Recovery Measures — Perioperative measures

SUMMARY:
ERAS IN TRAUMA Enhanced recovery after surgery (ERAS) or enhanced recovery protocols (ERP) is a concept first described by Kehlet in the early 1990s .Since its introduction, ERAS protocols have been successfully used in elective gastrointestinal surgery (colorectal, hepatobiliary and gastric), and there has been widespread acceptance and implementation in other surgical disciplines including urology, vascular , thoracic surgery and orthopaedics.

The approach employs a multimodal perioperative care pathway designed to attenuate the surgical stress response and accelerate postoperative recovery .

These benefits should be easily transferrable to the trauma patient population, if not greater, since trauma patients are generally younger, fitter and metabolically stable.

Trauma centres in developing countries constantly battle with reduced bed availability and restricted health care budgets. Optimization of health care practice is therefore urgent, particularly in trauma surgery.

Penetrating abdominal trauma is a major cause of morbidity and mortality in large urban trauma centres. It accounts for a significant number of hospital admissions and consumes a large portion of the health care budget.

In the trauma patient, the aim is to maintain the 'pre- injury' physiological status. Improving patient outcomes with reduced morbidity and early hospital discharge reduces the cost of treating these patients .

The small pilot study by Moydien et al., showed that ERPS can be successfully implemented with significant shorter hospital stays without any increase in postoperative complications in a select group of trauma patients undergoing emergency laparotomy for isolated penetrating abdominal trauma. Furthermore, the study showed that ERPS can also be applied to patients undergoing emergency surgery. Given the fact that penetrating abdominal trauma remains a substantial burden of disease, especially in developing countries such as South Africa, this proven approach to patient care in elective surgery can now be safely employed in the trauma and emergency setting.

Penetrating abdominal trauma remains a substantial burden of disease, especially in developing countries such as South Africa, and especially the Western Cape, where we have seen an increase in the number of trauma patients being treated for penetrating injuries at our level 1 centre. This has in turn led to severe constraints on the available resources, with the trauma ward often at maximum capacity with delayed discharges due to poor ambulation, post operative complications, and delay in return to enteral feeding.

Currently there is no randomized controlled study in the trauma literature, evaluating enhanced recovery after trauma procedures .It is our hypothesis to that implementing an "ERATS" protocol , will lead to a reduction in morbidity, reduction in hospital stay , with a subsequent decrease in costs. This will allow us to implement this as a new standard protocol , and thus change the current practice in stable penetrating trauma patients undergoing explorative laparotomy in our unit, nationally and worldwide.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* Penetrating abdominal trauma
* Require emergency laparotomy
* Alert ( Glasgow Coma Scale - 15/15)
* Able to consent
* Hemodynamically stable

Exclusion Criteria:

* Additional extra-abdominal injuries
* Spinal cord injuries
* Requiring damage control surgery from initial assessment (hemodynamically unstable )
* Do not consent to the study
* Need for ICU admission from initial surgery
* Pregnant patients
* All Duodenal injuries
* All Bladder injuries
* Previous laparotomies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | 7 days
  Duration of admission to the hospital

SECONDARY OUTCOMES:
Early feeding post explorative laparotomy | 7 days
  Days to tolerating full ward diet
Early removal of Nasogastric tubes, urinary catheters ,drains | 7 days
  Days to complete ambulation
Comparative mortality between the control and ERATS group | 30 days
  30 day mortality
Local aneasthetic wound infusion catheter system inserted in the laparotomy wound post procedure compared to standard opiate intravenous infusions used post operatively | 7 days
  Comparative daily pain score evaluation with Visual Analogue Score between control and ERATS group
Benefit of early mobilization post exploratory laparotomy | 7 days
  Time taken to return to normal activities of daily living, complete ambulation
Cost comparative between the 2 groups | 30 days
  Average cost between the 2 groups based on days in hospital , medication and consumables used
Morbidity in control group compared to ERATS group | 30 days
  Post operative surgical complications will be graded according to the extended Clavien-Dindo scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Nicol, FCS(SA), Study Director — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Vape, South Africa

IPD SHARING:
Plan to Share IPD: No